CLINICAL TRIAL: NCT03762603
Title: Does Supplementing of Quadriceps Strength With Exoskeleton After Total Knee Arthroplasty in High Risk Population Reduce Transfer to Extended Care Facility (ECF)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Derek Amanatullah, Assistant professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 45810
Record Dates: First submitted 2018-08-09; First posted 2018-12-04 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2022-05

CONDITIONS: Primary Knee Replacement Surgery
Keywords: Pneumatic; exoskeleton
MeSH Terms: interventions — Exoskeleton Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- robotic exoskeleton device (Experimental): Patients who are scheduled to be discharged to a ECF will be asked if they would want to use the exoskeleton device ( for which safety and comfort has been established) instead of going for ECF.
  Interventions: Device: Robotic exoskeleton device

INTERVENTIONS:
Device: Robotic exoskeleton device — It is a non invasive and non significant risk medical device which wraps around operated knee to support motion.

SUMMARY:
This study involves an exoskeleton which is believed to increase quadriceps muscle strength in the rehabilitation phase after TKA and reduce the discharge the such patients in Extended care facility (ECF) . The purpose of this study is to access efficacy of the robotic exoskeleton device wrapped around the operated knee on patients

ELIGIBILITY:
Inclusion criteria

1. Patients undergoing unilateral primary knee replacement surgery
2. Patients who pre-operatively desire discharged to ECF
3. Patients willing and capable to sign the written informed consent

Exclusion criteria

1. Patients undergoing bilateral primary knee replacement surgery
2. Patients undergoing revision knee replacement surgery
3. Patients who pre-operatively desire discharged to Home
4. Patients not willing and capable to sign the written informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Predicting discharge location after TKA | 2 years
  The objective of this study is to observe how many patients are not transferred to ECF in the post-surgery time period as a result of using a robotic exoskeleton on operated knee. We will list number of patients NOT going for ECF.

SECONDARY OUTCOMES:
Evaluate the effectiveness of the robotic exoskeleton device at time of discharge | upto 2 weeks
  To assess the effectiveness of the device by evaluating the number of patients discharge with exoskeleton device along with Home Health Services all by using questionnaire
Evaluate the effectiveness of the robotic exoskeleton device at time of discharge | upto 2 weeks
  We plan to determine patient length of stay in hospital ( in hours)
Evaluate the effectiveness of the robotic exoskeleton device at time of discharge | upto 2 weeks
  Determining patients performance of Stairs at discharge. Patients at the time of discharge are asked to step 3 stairs and answer related questions using a questionnaire
Evaluate the effectiveness of the robotic exoskeleton device at time of discharge through 2 years | up to 2 years
  To assess the effectiveness of the device by calculating Initial knee society score (KSS) and Knee society score at 2 weeks, 3 months and 2 years after surgery. The scale ranges from 0-100 with grading as Score 80-100 - Excellent Score 70-79 - Good Score 60-69 - Fair Score below 60 - Poor
Evaluate the effectiveness of the robotic exoskeleton device at time of discharge through 2 years | up to 2 years
  To assess the effectiveness of the device by calculating initial Range of motion ( ROM) at the time of discharge and at 2 weeks, 3 months and 2 years after surgery.
Evaluate the effectiveness of the robotic exoskeleton device at time of discharge through 2 years | up to 2 years
  To assess the effectiveness of the device by examining Gait Aide use at discharge, 2 weeks, 3 months and 2 years after surgery. This is done to examine performance . The gait aide use provident ranges as Nothing > Cane > crutch > walker
Evaluate the effectiveness of the robotic exoskeleton device at time of discharge through 2 years | up to 2 years
  calculating Timed-up-and-Go at discharge, 3 months and 2 years after surgery
Evaluate the effectiveness of the robotic exoskeleton device at post operative follow up | 2 weeks and 3 months
  calculating device compliance (on/off) at 2 weeks and 3 months after surgery using a questionnaire
Evaluate the effectiveness of the robotic exoskeleton device at post operative follow up | 2 weeks and 3 months
  To assess the effectiveness of device by calculating number of Falls at 2 weeks and 3 months using a questionnaire
Evaluate the effectiveness of the robotic exoskeleton device at post operative follow up | 2 weeks and 3 months
  To assess the effectiveness of device by calculating Initial satisfaction with the device and satisfaction at 2 weeks and 3 months after surgery using a questionnaire. The scale ranges from:
  Very satisfied Satisfied Neutral Not satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Derek Amanatullah, M.D. PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtz S, Mowat F, Ong K, Chan N, Lau E, Halpern M. Prevalence of primary and revision total hip and knee arthroplasty in the United States from 1990 through 2002. J Bone Joint Surg Am. 2005 Jul;87(7):1487-97. doi: 10.2106/JBJS.D.02441. PMID 15995115
- [Background] Losina E, Walensky RP, Kessler CL, Emrani PS, Reichmann WM, Wright EA, Holt HL, Solomon DH, Yelin E, Paltiel AD, Katz JN. Cost-effectiveness of total knee arthroplasty in the United States: patient risk and hospital volume. Arch Intern Med. 2009 Jun 22;169(12):1113-21; discussion 1121-2. doi: 10.1001/archinternmed.2009.136. PMID 19546411
- [Background] Healy WL, Rana AJ, Iorio R. Hospital economics of primary total knee arthroplasty at a teaching hospital. Clin Orthop Relat Res. 2011 Jan;469(1):87-94. doi: 10.1007/s11999-010-1486-2. PMID 20694537
- [Background] Schwarzkopf R, Ho J, Quinn JR, Snir N, Mukamel D. Factors Influencing Discharge Destination After Total Knee Arthroplasty: A Database Analysis. Geriatr Orthop Surg Rehabil. 2016 Jun;7(2):95-9. doi: 10.1177/2151458516645635. Epub 2016 Apr 26. PMID 27239383
- [Background] Goto K, Morishita T, Kamada S, Saita K, Fukuda H, Shiota E, Sankai Y, Inoue T. Feasibility of rehabilitation using the single-joint hybrid assistive limb to facilitate early recovery following total knee arthroplasty: A pilot study. Assist Technol. 2017 Winter;29(4):197-201. doi: 10.1080/10400435.2016.1219883. Epub 2016 Aug 10. PMID 27689789